CLINICAL TRIAL: NCT03780530
Title: Comparison of Different Techniques for Perineal Skin Closure During Mediolateral Episiotomy Repair
Brief Title: Different Techniques for Perineal Skin Closure During Mediolateral Episiotomy Repair
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Radwa Rasheedy Ali, Principal Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ain shams maternity U
Record Dates: First submitted 2018-12-16; First posted 2018-12-19 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Episiotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- subcuticular suturing (Active Comparator)
  Interventions: Procedure: subcuticular suturing
- surgical glue (Active Comparator)
  Interventions: Procedure: Surgical glue
- adhesive steri-strip tape (Active Comparator)
  Interventions: Procedure: adhesive steri-strip tape

INTERVENTIONS:
Procedure: subcuticular suturing — Those undergoing Subcuticular suturing of perineal skin using 910 polyglactin vicryl No 2/0 (EGYCRYL®).
  Arms: subcuticular suturing
Procedure: Surgical glue — Those undergoing perineal skin closure using adhesive glue n-butyl-2-cyanoacrylate (Histoacryl®).
  Arms: surgical glue
Procedure: adhesive steri-strip tape — Those undergoing closure of perineal skin via Adhesive surgical water-resistant tape application. (3M® Transpore™ Surgical Tapes).
  Arms: adhesive steri-strip tape

SUMMARY:
this study aims to assess the efficacy and the safety of various cosmetic techniques (subcuticular, surgical glue, adhesive tapes) for perineal skin closure during mediolateral episiotomy repair

ELIGIBILITY:
Inclusion Criteria:

* Women aged above 18 yrs.
* Primiparous.
* Undergoing spontaneous vaginal delivery of a single full-term fetus.
* Vertex presentation.
* Having mediolateral episiotomy.

Exclusion Criteria:

* Body mass index ≥ 35 kg/m2
* Complicated delivery by any tears other than episiotomy or postpartum hemorrhage.
* Any risk factor causing increased stretch of the perineum; Operative vaginal delivery, fetal macrosomia.
* The use of epidural anesthesia.
* Previous perineal surgeries, local infection or lesions.
* Any medical condition that can cause excessive bleeding or impair wound healing; (cardiovascular disease, diabetes, anemia, coagulopathy, collagen disease or Immunosuppression).
* Contraindication or Hypersensitivity to any of materials used in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2019-10-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Short -term postpartum pain | six hours postpartum
  Post-operative perineal pain will be evaluated at 6 hrs after the procedure using visual analogue scale patient to choose a number from 0 to 10 that best describes their current pain. 0 would mean "no pain" and 10 would mean "worst possible pain
Short -term postpartum pain | 10 days postnatal
  Post-operative perineal pain will be evaluated at 10 days after the procedure using visual analogue scale patient to choose a number from 0 to 10 that best describes their current pain. 0 would mean "no pain" and 10 would mean "worst possible pain